CLINICAL TRIAL: NCT04419987
Title: Study of the Functionality of New Genetic Variants at the Origin of Constitutional Platelet Disease.
Brief Title: Study of Constitutional Platelet Disease
Acronym: EVGPP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-30
Record Dates: First submitted 2020-05-03; First posted 2020-06-09 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-04

CONDITIONS: Blood Platelet Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- constitutional platelet patholog (Experimental): Patient and relatives having a constitutional platelet pathology
  Interventions: Genetic: draw blood

INTERVENTIONS:
Genetic: draw blood — search for new genetic variations (when the diagnostic exploration will have been non informative) by sequencing exons.

SUMMARY:
Platelets are circulating blood cells. They bind to each other and to the wall of the damaged vessel to prevent excessive blood loss.

Platelets can be :

* insufficient in number in the case of thrombocytopenia;
* or non-functional in the case of thrombopathy. Constitutional thrombopathies and thrombopenias are rare diseases. Constitutional thrombopenias cause haemorrhage of variable intensity and are sometimes a sign of more serious haematological pathologies. The evolutionary risk of some constitutional thrombopenias is the appearance of myelofibrosis, dysmyelopoiesis or malignant proliferation. While the evolutionary stakes of some thrombopenias and especially syndromic thrombopenias will be more likely to affect other organs (kidney, heart, bones, brain, ...), other constitutional thrombopenias will have few consequences. Their diagnosis will then have the major challenge of distinguishing them from immunological thrombopenias and avoiding the use of inappropriate and sometimes severe treatments (corticosteroids, IV immunoglobulins, immunosuppressants, splenectomy). Mutations in more than forty genes have been identified to date and are responsible for thrombocytopenia.

Constitutional thrombopathies are heterogeneous and may involve different platelet constituents. In short, when platelets are stimulated at a lesion site, various soluble or matrix agonists bind to platelet receptors to induce calcium flow, secretion and platelet aggregation at a vascular gap to prevent blood loss. Constitutional thrombopathies are primarily at risk of spontaneous or induced mucocutaneous bleeding. Some thrombopathies are also part of more complex syndromic patterns. In recent decades, considerable progress has been made in the understanding of thrombopathies, enabling them to be better identified. Details have been provided on platelet dysfunctions linked to abnormalities in the processes of granule biogenesis and secretion, and to signalling defects (in particular surface receptor deficiency). Currently, more than thirty genes are the site of autosomal dominant, recessive or X-linked mutations and can be sequenced.

DETAILED DESCRIPTION:
Platelets are circulating blood cells. They bind to each other and to the wall of the damaged vessel to prevent excessive blood loss.

Platelets can be :

* insufficient in number in the case of thrombocytopenia;
* or non-functional in the case of thrombopathy. Constitutional thrombopathies and thrombopenias are rare diseases. Constitutional thrombopenias cause haemorrhage of variable intensity and are sometimes a sign of more serious haematological pathologies. The evolutionary risk of some constitutional thrombopenias is the appearance of myelofibrosis, dysmyelopoiesis or malignant proliferation. While the evolutionary stakes of some thrombopenias and especially syndromic thrombopenias will be more likely to affect other organs (kidney, heart, bones, brain, ...), other constitutional thrombopenias will have few consequences. Their diagnosis will then have the major challenge of distinguishing them from immunological thrombopenias and avoiding the use of inappropriate and sometimes severe treatments (corticosteroids, IV immunoglobulins, immunosuppressants, splenectomy). Mutations in more than forty genes have been identified to date and are responsible for thrombocytopenia.

Constitutional thrombopathies are heterogeneous and may involve different platelet constituents. In short, when platelets are stimulated at a lesion site, various soluble or matrix agonists bind to platelet receptors to induce calcium flow, secretion and platelet aggregation at a vascular gap to prevent blood loss. Constitutional thrombopathies are primarily at risk of spontaneous or induced mucocutaneous bleeding. Some thrombopathies are also part of more complex syndromic patterns. In recent decades, considerable progress has been made in the understanding of thrombopathies, enabling them to be better identified. Details have been provided on platelet dysfunctions linked to abnormalities in the processes of granule biogenesis and secretion, and to signalling defects (in particular surface receptor deficiency). Currently, more than thirty genes are the site of autosomal dominant, recessive or X-linked mutations and can be sequenced.

A national organisation has been set up for the molecular diagnosis of these pathologies. DNA samples from patients meeting strict criteria (familial nature, chronic pathology, associated signs) are sent to the molecular biology departments. A panel of 80 genes is then sequenced in order to identify genetic variations potentially responsible for the pathology. In 40% of cases, a diagnosis of certainty will be made. For the remaining 60%, the analysis will remain non-informative for several reasons:

* Either it is a question of revealing a variation in a known gene but not yet described in the literature, the deleterious nature of which must be confirmed;
* or no gene has been identified and there will be an indication of a broader sequencing involving all exons in the genome. This strategy has already enabled the coordinating site to identify several new genes of particular importance;
* either they are individuals for which the constitutional character was not sufficiently documented, a diagnostic reorientation will then be necessary.

This project will consist of proving the deleterious nature of new genetic variations using cellular and molecular biology methods. These variations will be either those identified on a known gene in the context of diagnosis (sequencing of a panel of genes) or those identified by sequencing exons on a gene not yet known to be involved in constitutional platelet pathologies. The sequencing of exons is an integral part of the project.

ELIGIBILITY:
Inclusion Criteria:

* Adult or minor over 7 years old.
* Patient and relatives with a constitutional platelet pathology (familial thrombocytopenia resulting in a platelet count < 150 G.L-1 in several family members and/or familial thrombopathy resulting in platelet dysfunction in several members of a family) for which a genetic variation has been demonstrated but whose deleterious nature remains to be confirmed.
* Patient and relatives having a constitutional platelet pathology (familial thrombocytopenia resulting in a platelet count < 150 G.L-1 in several members of the family and/or familial thrombopathy resulting in platelet dysfunction in several members of a family) for which the genetic diagnosis has not revealed any variation potentially implicated in the pathology.

Exclusion Criteria:

* Minor under 7 years of age.
* Patient with no platelet pathology.
* Patient with platelet disease: non-chronic, non-familial.
* Patient with a familial platelet disease with a known deleterious mutation.obviously acquired.

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2020-07-20 (Estimated); Primary Completion 2020-12-20 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Adhesion | 5 years
  Isolated wafers are deposited on substrate coated plates, the wafers adhere to the substrate. Then the number of adherent wafers will be counted by cell imaging. Several substrates will be tested.
Study of platelet protein expression | 5 years
  A western blot will be made from the platelet lysate, allowing the detection of specific proteins with the help of antibodies directed against the proteins of interest.
  A semi-quantitative analysis of these proteins will be performed by chemiluminescence.